CLINICAL TRIAL: NCT02998125
Title: A Psychometric Analysis of the Arabic Version of Oxford Knee Score Before and After Total Knee Arthroplasty in a Middle East Population and an Exploration of Outcomes Post-total Knee Arthroplasty in the Middle East
Brief Title: An Exploration of Outcomes Post-total Knee Arthroplasty in Middle East
Status: Completed | Type: Observational
Sponsor: University of Salford (Other)
Collaborators: King Khalid University Hospital (Other); Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Bodor Bin sheeha, PhD student at University of Salford, University of Salford
Other Study IDs: USalford-Bsheeha
Record Dates: First submitted 2016-12-14; First posted 2016-12-20 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- before and after total knee arthroplasty: assess the functional outcome before and 6 months after total knee arthroplasty
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — prospective assessments for the functional outcome before and after the total knee arthroplasty

SUMMARY:
The intention is to explore whether there are factors, which can help us to understand why some patient outcomes, following total knee arthroplasty are not successful and identify prediction factors for progression. Assessment of outcomes pre- and post-surgery with objective tools is a way to explore prediction tools for good/poor progression and improve patient selection and timing for surgery.

The first aim of this project is determine the psychometric properties of the Arabic Version of Oxford Knee Score, including internal consistency, reliability and validity before and post-total knee arthroplasty in both males and females in a Middle East population. The second aim is to assess the reliability of the Star Excursion Balance Test for measuring the dynamic balance. The final aim is explore outcomes post-total knee arthroplasty among Middle East patients using the Arabic Version of Oxford Knee Score, physical activity measures and performance-based measurements such as: 30 s chair-stand test, stair-climb test, timed up-and-go test and a 6 m walk test while adhering to Osteoarthritis Research Society International recommendations.

DETAILED DESCRIPTION:
Project objectives

To gain an understanding of recovery post-TKA in a Saudi population and explore whether there are factors which can help us to understand why some patient outcomes are not successful and identify prediction factors for progression. It is a prospective study measuring outcomes six months post-TKA with the following objectives:

* Examine the internal consistency, reliability and validity of the Arabic Version of Oxford Knee Score before and after total knee arthroplasty in both male and female Middle East patients.
* Examine the test- re-test reliability of the Star Excursion Balance Test in both male and female Middle Eastern patients.
* Measure patient outcomes post-total knee arthroplasty using patient self-reporting activity measurements and the Arabic Version of Oxford Knee Score;
* Evaluate physical activity level improvements post-knee arthroplasty using objective methods and an accelerometer: ActivPAL;
* Assess functional recovery post-knee arthroplasty according to Osteoarthritis Research Society International recommendations using performance-based measurements, such as: 30 s chair-stand test, stair-climb test, timed up-and-go test and a 6 m walk test alongside functional balance.

The rationale which led to this project;

Knee osteoarthritis (OA) is a major cause of disability around the world; it is the most common chronic condition in primary care in the UK. By 2030 it is predicted to be the greatest cause of disability in the general population . An effective end-stage treatment for knee OA is knee-replacement surgery, which was first done in the 1970s and 1980s.

In England and Wales, the number of knee-replacement procedures recorded by the National Joint Registry in 2013 was 91,703, which represents an increase of 0.9 % over 2012. The data analysis by the National Joint Registry and the Office of National Statistics suggests that, by 2030, primary TKAs will increase by 117% from the 2012 level. Subsequently, TKA revision surgeries are expected to increase incrementally by 332%. There is a similar estimation of demand for revision TKA surgeries in the United States; by 2030, they are expected to rise by 601% from the 2005 level. The United States estimation of primary TKA is for growth of 673% from the 2005 level, which is similar to England and Wales's upper-limit projections.

Post-TKA, 75-85% of patients report satisfaction with surgery outcomes, while the remaining 15-25% are dissatisfied (Klit, Jacobsen, Rosenlund, Sonne-Holm, & Troelsen, 2014). Total knee arthroplasty's success has traditionally been evaluated from the surgeon's perspective, e.g. the presence of surgical complications or implant survival. This is gradually changing to involve the patient in measuring health outcomes and decision-making processes. Patient-reported outcome measures (PROMs) have evolved to explore patient perspectives by monitoring the quality of care in health organizations and conducting clinical trial outcomes.

PROM results cannot exclude the Research Participant Effect (RPE) or subjective over/underestimation due to psychosocial effects or pain from other joints, such as hips or back. Hence, objective clinical evaluation methods can minimize patients' subjective over/underestimations of outcomes, though RPE can not be excluded. Objective assessment has some advantages over PROMs, such as a lack of ceiling effects and more precision and responsiveness, and it does not require cultural and language adaptation. Performance-based Outcome Measures (PBOMs) have the advantage of being objective measures that do not overlap with pain measurement. They are sensitive to detecting change, responsive, have a minimal ceiling effect and are feasible.

PROMs and PBOM measurement tools assess different aspects of function post-TKA. PROMs mainly assess patients' functional ability beliefs and experiences, while objective functional assessment instruments and PBOM measurement tools evaluate patients' actual ability and function. Therefore, to conduct comprehensive functional assessments post-TKA, PROMs, objective functional assessment instruments and PBM measurement tools are recommended.

To the best of our knowledge, no study has explored the outcome post TKA using the PROMs, PBOMs and functional balance measurement tools in Saudi male and female population or explored possible accurate prediction factors for outcomes post-TKA. Reliable outcome prediction could, however, improve patient selection for surgery, as appropriate timing for surgery depends on patient symptoms and efficient patient preparation for surgery if it is to be cost-effective. Accurate preoperative prediction is crucial to minimize the potential for unrealistic expectations about outcomes.

This study will investigate outcomes post-total knee arthroplasty and factors that may predict good/poor progression using three categories of outcome measurements in order to minimize subjective over/ underestimation of surgical outcomes. Thus, the study seeks to explore accurate and objective prediction factors of post-total knee arthroplasty progression.

Potentially, reliable outcome predictions could improve patient selection for surgery, as appropriate timing for surgery depends on patients' symptoms and efficient patient preparation for surgery, if it is to be cost-effective. Accurate preoperative prediction is crucial to minimize the potential for unrealistic expectations about outcomes.

ELIGIBILITY:
Inclusion Criteria:

All patients will be asked to participate during preadmission orthopedics clinic visits to King Khalid University Hospital in Riyadh if the patient;

* Scheduled for elective primary unilateral total knee arthroplasty.
* For end-stage knee osteoarthritis.
* In a stable and controlled medical condition,

Exclusion Criteria:

* Are scheduled for bilateral knee arthroplasty or unilateral knee revision surgery;
* Cannot read and understand Arabic
* Have limited function due to musculoskeletal conditions other than unilateral knee osteoarthritis.
* Have been diagnosed with uncontrolled diabetes mellitus or blood pressure.
* Have been diagnosed with any neurologic disorders, such as stroke, Parkinson's disease or multiple sclerosis.
* Are morbidly obese and have a body mass index (BMI) greater than 40.
* Have advance osteoporosis or some other unstable chronic disease.
* Have been diagnosed with a peripheral vascular or uncontrolled cardiac disease.
* Participant will further be excluded post-surgery if they develop any surgical complications, such as deep vein thrombosis, uncontrolled infection or fracture.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The present study is a prospective six and twelve month follow-up trial to explore the outcome post TKA in addition to assess the validity, reliability and responsiveness of the Arabic version of Oxford Knee Score and the Star Excursion Balance Test with total knee arthroplasty patients.
  An information sheet will be given to all participants who agree to participate to clarify the objectives of the study. Before participating, patients will need to sign a consent form (Appendix 2) and they will have the right to clarify any concerns about the study with the researcher. A patient's participation or otherwise will not affect the quality of service, all patients will receive conventional orthopedic care and a standard level of physiotherapy according to hospital protocols.
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Performance based measurements change in Thirty second chair-stand test | one week before admission day and 6 months after surgery to assess the performance changes post-surgery
  A chair of 17 inches (45cm) height is used as the starting position for patients sitting with their arms cross the chest. Patients are instructed to stand and then sit with good buttock placement and back support, their hands on arm rests and feet correctly placed, then stand again as fast and safely as they can. The assessor counts the number of complete chair stands within 30 s. The mean of two trials will be used for analysis (Gill & McBurney, 2008; Unver, Kalkan, Yuksel, Kahraman, & Karatosun, 2015)
Performance based measurements change in Stair-climb test | one week before admission day and 6 months after surgery to assess the performance changes post-surgery
  Using a stopwatch accurate to 1/100 s, an assessor will measure the time required for a patient, using a handrail if required, to ascend and descend a flight of twelve steps 18 cm high and 28 cm deep. Patients will be instructed to ascend and descend the stairs as quickly, safely and comfortably as they can. The mean of two trials will be used for analysis (Mizner et al., 2011)
Performance based measurements change in Timed up-and-go test | one week before admission day and 6 months after surgery to assess the performance changes post-surgery
  The test procedure will use a stopwatch accurate to 1/100 s; a chair of standard 45 cm height, with armrests, will be placed on an outdoor level footpath and a line 3 metres from the chair will be drawn. Patients will be instructed to stand up from the chair, using the arms if required, walk for 3 metres to the line, then turn round and walk to sit back down on the chair as quickly, safely and comfortably as they can. An assessor will start timing as the patient leans forward to stand up, and stop when the patient's hips make contact with the seat to sit down. An average of two repetitions will be analysed (Ko, Naylor, Harris, Crosbie, & Yeo, 2013; Mizner et al., 2011; Podsiadlo & Richardson, 1991).
Performance based measurements change in Six minute walk test | one week before admission day and 6 months after surgery to assess the performance changes post-surgery
  The test will measure how far patients can walk in 6 minutes along a level 25-metre footpath. Patients can use an assistive device if required, take a rest if necessary and have standardized encouragement after each minute. The assessor will ask the patient to stop after 6 minutes. Only one test will be performed to avoid fatigue ("ATS Statement," 2002; Ko et al., 2013; Mizner et al., 2011).
Balance change | one week before admission day and 6 months after surgery to assess the balance changes post-surgery
  In the Star Excursion Balance Test, three tape measures will be fixed to the clinic floor, one oriented anteriorly to the apex and two aligned at 135° to the anterior tape in the posterolateral and posteromedial directions. (Fullam, Caulfield, Coughlan, & Delahunt, 2014).
  The patient will stand in the center of the grid and be instructed to stand on the affected or operated leg while reaching out as far as possible in one of the three directions with the other lower extremity, and then return that leg to the center. The participant will be asked to perform the test barefoot, keeping the heel of the stance leg on the floor at all times and to bend the knee of the stance leg. If the participant does not carry out any of these instructions, the trial will repeated.
  The assessor will measure the reach distance in each direction in centimeters and then normalize the average of the three trials to leg length.
Physical activity measurements change will be assess using an activPAL activity monitor (PAL Technologies, Glasgow, UK) | one week before admission day and 6 months after surgery to assess the physical activity changes post-surgery
  an activPAL activity monitor (PAL Technologies, Glasgow, UK) as this proven accelerometer provides objective quantification of free-living physical activity without any modification (Dahlgren, Carlsson, Moorhead, Hager-Ross, & McDonough, 2010; Schmalzried et al., 1998). It is suitable as it light in weight (20g), includes an inclinometer and is small in size (53 x 35 x 7 mm) Figure 3. The device is worn by patient's mid-thigh, secured by non-allergic waterproof adhesive tape under their clothes, for 7-10 days before surgery and 6 months after. Clear written and verbal instructions will be given to patients as they have to wear it all day and all night except, when bathing or swimming (they can take a shower with it on).

SECONDARY OUTCOMES:
Arabic versions of Oxford Knee Score Validity assessment | one week before admission day
  The patients will be instructed to complete the Arabic versions of Oxford Knee Score, Arabic versions of Knee injury and Osteoarthritis Outcome Score (KOOS) and visual analogue scale (VAS) before Arthroplasty as baseline data in order to assess the correlation of Arabic versions of Oxford Knee Score with the Arabic version of KOOS and VAS to determine construct validity (Arabic versions of Oxford Knee Score, Knee injury and Osteoarthritis Outcome Score and visual analogue scale
Arabic versions of Oxford Knee Score Reliability assessment | one week before admission day, admission day and 6 months after surgery and to evaluate the construct validity of the Arabic version of Oxford Knee Score
  Patients will be asked to fill out Arabic forms independently without any interpretation to assess the Score reliability and responsiveness.

CONTACTS AND LOCATIONS:
Locations (1):
- King Khalid University Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Bade MJ, Kohrt WM, Stevens-Lapsley JE. Outcomes before and after total knee arthroplasty compared to healthy adults. J Orthop Sports Phys Ther. 2010 Sep;40(9):559-67. doi: 10.2519/jospt.2010.3317. PMID 20710093
- [Background] Bade MJ, Wolfe P, Zeni JA, Stevens-Lapsley JE, Snyder-Mackler L. Predicting poor physical performance after total knee arthroplasty. J Orthop Res. 2012 Nov;30(11):1805-10. doi: 10.1002/jor.22140. Epub 2012 Apr 26. PMID 22539338
- [Background] Bullens PH, van Loon CJ, de Waal Malefijt MC, Laan RF, Veth RP. Patient satisfaction after total knee arthroplasty: a comparison between subjective and objective outcome assessments. J Arthroplasty. 2001 Sep;16(6):740-7. doi: 10.1054/arth.2001.23922. PMID 11547372
- [Background] Carr AJ, Robertsson O, Graves S, Price AJ, Arden NK, Judge A, Beard DJ. Knee replacement. Lancet. 2012 Apr 7;379(9823):1331-40. doi: 10.1016/S0140-6736(11)60752-6. Epub 2012 Mar 6. PMID 22398175
- [Background] Charoencholvanich K, Pongcharoen B. Oxford knee score and SF-36: translation & reliability for use with total knee arthroscopy patients in Thailand. J Med Assoc Thai. 2005 Sep;88(9):1194-202. PMID 16536104
- [Background] Coughlan GF, Fullam K, Delahunt E, Gissane C, Caulfield BM. A comparison between performance on selected directions of the star excursion balance test and the Y balance test. J Athl Train. 2012 Jul-Aug;47(4):366-71. doi: 10.4085/1062-6050-47.4.03. PMID 22889651
- [Background] Dahlgren G, Carlsson D, Moorhead A, Hager-Ross C, McDonough SM. Test-retest reliability of step counts with the ActivPAL device in common daily activities. Gait Posture. 2010 Jul;32(3):386-90. doi: 10.1016/j.gaitpost.2010.06.022. Epub 2010 Jul 22. PMID 20655228
- [Background] Dobson F, Hinman RS, Roos EM, Abbott JH, Stratford P, Davis AM, Buchbinder R, Snyder-Mackler L, Henrotin Y, Thumboo J, Hansen P, Bennell KL. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. Osteoarthritis Cartilage. 2013 Aug;21(8):1042-52. doi: 10.1016/j.joca.2013.05.002. Epub 2013 May 13. PMID 23680877
- [Background] Field, A. (2009). Discovering Statistics Using SPSS: SAGE Publications Ltd,.
- [Background] Fullam K, Caulfield B, Coughlan GF, Delahunt E. Kinematic analysis of selected reach directions of the Star Excursion Balance Test compared with the Y-Balance Test. J Sport Rehabil. 2014 Feb;23(1):27-35. doi: 10.1123/jsr.2012-0114. Epub 2013 Aug 12. PMID 23945793
- [Background] Gill S, McBurney H. Reliability of performance-based measures in people awaiting joint replacement surgery of the hip or knee. Physiother Res Int. 2008 Sep;13(3):141-52. doi: 10.1002/pri.411. PMID 18697226
- [Background] Gribble PA, Hertel J, Plisky P. Using the Star Excursion Balance Test to assess dynamic postural-control deficits and outcomes in lower extremity injury: a literature and systematic review. J Athl Train. 2012 May-Jun;47(3):339-57. doi: 10.4085/1062-6050-47.3.08. PMID 22892416
- [Background] Harris K, Dawson J, Doll H, Field RE, Murray DW, Fitzpatrick R, Jenkinson C, Price AJ, Beard DJ. Can pain and function be distinguished in the Oxford Knee Score in a meaningful way? An exploratory and confirmatory factor analysis. Qual Life Res. 2013 Nov;22(9):2561-8. doi: 10.1007/s11136-013-0393-x. Epub 2013 Mar 23. PMID 23526094
- [Background] Hertel J, Braham RA, Hale SA, Olmsted-Kramer LC. Simplifying the star excursion balance test: analyses of subjects with and without chronic ankle instability. J Orthop Sports Phys Ther. 2006 Mar;36(3):131-7. doi: 10.2519/jospt.2006.36.3.131. PMID 16596889
- [Background] Hossain FS, Konan S, Patel S, Rodriguez-Merchan EC, Haddad FS. The assessment of outcome after total knee arthroplasty: are we there yet? Bone Joint J. 2015 Jan;97-B(1):3-9. doi: 10.1302/0301-620X.97B1.34434. PMID 25568406
- [Background] Hossain FS, Patel S, Fernandez MA, Konan S, Haddad FS. A performance based patient outcome score for active patients following total knee arthroplasty. Osteoarthritis Cartilage. 2013 Jan;21(1):51-9. doi: 10.1016/j.joca.2012.09.019. Epub 2012 Oct 9. PMID 23063619
- [Background] Hyong IH, Kim JH. Test of intrarater and interrater reliability for the star excursion balance test. J Phys Ther Sci. 2014 Aug;26(8):1139-41. doi: 10.1589/jpts.26.1139. Epub 2014 Aug 30. PMID 25202168
- [Background] Impellizzeri FM, Mannion AF, Leunig M, Bizzini M, Naal FD. Comparison of the reliability, responsiveness, and construct validity of 4 different questionnaires for evaluating outcomes after total knee arthroplasty. J Arthroplasty. 2011 Sep;26(6):861-9. doi: 10.1016/j.arth.2010.07.027. Epub 2010 Nov 12. PMID 21074964
- [Background] Jagger, C., Matthews, R., Spiers, N., Brayne, C., Comas - Herrera, A., Robinson, T., . . . Croft, P. (2006). Compression or expansion of disability?: forecasting future disability levels under changing patterns of diseases: King's Fund.
- [Background] Jenny JY, Diesinger Y. Validation of a French version of the Oxford knee questionnaire. Orthop Traumatol Surg Res. 2011 May;97(3):267-71. doi: 10.1016/j.otsr.2010.07.009. Epub 2011 Jan 12. PMID 21233035
- [Background] Kennedy DM, Stratford PW, Wessel J, Gollish JD, Penney D. Assessing stability and change of four performance measures: a longitudinal study evaluating outcome following total hip and knee arthroplasty. BMC Musculoskelet Disord. 2005 Jan 28;6:3. doi: 10.1186/1471-2474-6-3. PMID 15679884
- [Background] Klit J, Jacobsen S, Rosenlund S, Sonne-Holm S, Troelsen A. Total knee arthroplasty in younger patients evaluated by alternative outcome measures. J Arthroplasty. 2014 May;29(5):912-7. doi: 10.1016/j.arth.2013.09.035. Epub 2013 Oct 1. PMID 24269097
- [Background] Ko V, Naylor JM, Harris IA, Crosbie J, Yeo AE. The six-minute walk test is an excellent predictor of functional ambulation after total knee arthroplasty. BMC Musculoskelet Disord. 2013 Apr 24;14:145. doi: 10.1186/1471-2474-14-145. PMID 23617377
- [Background] Lungu E, Desmeules F, Dionne CE, Belzile EL, Vendittoli PA. Prediction of poor outcomes six months following total knee arthroplasty in patients awaiting surgery. BMC Musculoskelet Disord. 2014 Sep 8;15:299. doi: 10.1186/1471-2474-15-299. PMID 25201448
- [Background] Lutzner C, Kirschner S, Lutzner J. Patient activity after TKA depends on patient-specific parameters. Clin Orthop Relat Res. 2014 Dec;472(12):3933-40. doi: 10.1007/s11999-014-3813-5. Epub 2014 Jul 23. PMID 25053290
- [Background] McCambridge J, Witton J, Elbourne DR. Systematic review of the Hawthorne effect: new concepts are needed to study research participation effects. J Clin Epidemiol. 2014 Mar;67(3):267-77. doi: 10.1016/j.jclinepi.2013.08.015. Epub 2013 Nov 22. PMID 24275499
- [Background] Meiring RM, Frimpong E, Mokete L, Pietrzak J, Van Der Jagt D, Tikly M, McVeigh JA. Rationale, design and protocol of a longitudinal study assessing the effect of total knee arthroplasty on habitual physical activity and sedentary behavior in adults with osteoarthritis. BMC Musculoskelet Disord. 2016 Jul 13;17:281. doi: 10.1186/s12891-016-1141-5. PMID 27411316
- [Background] Mizner RL, Petterson SC, Clements KE, Zeni JA Jr, Irrgang JJ, Snyder-Mackler L. Measuring functional improvement after total knee arthroplasty requires both performance-based and patient-report assessments: a longitudinal analysis of outcomes. J Arthroplasty. 2011 Aug;26(5):728-37. doi: 10.1016/j.arth.2010.06.004. Epub 2010 Sep 20. PMID 20851566
- [Background] Naal FD, Impellizzeri FM, Sieverding M, Loibl M, von Knoch F, Mannion AF, Leunig M, Munzinger U. The 12-item Oxford Knee Score: cross-cultural adaptation into German and assessment of its psychometric properties in patients with osteoarthritis of the knee. Osteoarthritis Cartilage. 2009 Jan;17(1):49-52. doi: 10.1016/j.joca.2008.05.017. Epub 2008 Jul 7. PMID 18602843
- [Background] Palmer CR. Encyclopedia of biostatistics. BMJ. 1999 Feb 20;318(7182):542. doi: 10.1136/bmj.318.7182.542. No abstract available. PMID 10024284
- [Background] Patel A, Pavlou G, Mujica-Mota RE, Toms AD. The epidemiology of revision total knee and hip arthroplasty in England and Wales: a comparative analysis with projections for the United States. A study using the National Joint Registry dataset. Bone Joint J. 2015 Aug;97-B(8):1076-81. doi: 10.1302/0301-620X.97B8.35170. PMID 26224824
- [Background] Plichta, S., & Kelvin, E. (2012). Munro's Statistical Methods for Health Care Research: Lippincott Williams & Wilkins.
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Robinson RH, Gribble PA. Support for a reduction in the number of trials needed for the star excursion balance test. Arch Phys Med Rehabil. 2008 Feb;89(2):364-70. doi: 10.1016/j.apmr.2007.08.139. PMID 18226664
- [Background] Schmalzried TP, Szuszczewicz ES, Northfield MR, Akizuki KH, Frankel RE, Belcher G, Amstutz HC. Quantitative assessment of walking activity after total hip or knee replacement. J Bone Joint Surg Am. 1998 Jan;80(1):54-9. PMID 9469309
- [Background] Stratford PW, Kennedy DM. Performance measures were necessary to obtain a complete picture of osteoarthritic patients. J Clin Epidemiol. 2006 Feb;59(2):160-7. doi: 10.1016/j.jclinepi.2005.07.012. Epub 2005 Dec 27. PMID 16426951
- [Background] Thumboo J, Chew LH, Lewin-Koh SC. Socioeconomic and psychosocial factors influence pain or physical function in Asian patients with knee or hip osteoarthritis. Ann Rheum Dis. 2002 Nov;61(11):1017-20. doi: 10.1136/ard.61.11.1017. PMID 12379527
- [Background] Unver B, Kalkan S, Yuksel E, Kahraman T, Karatosun V. Reliability of the 50-foot walk test and 30-sec chair stand test in total knee arthroplasty. Acta Ortop Bras. 2015 Jul-Aug;23(4):184-7. doi: 10.1590/1413-78522015230401018. PMID 26327798